CLINICAL TRIAL: NCT03065244
Title: KIDCARE (Kawasaki Disease Comparative Effectiveness Trial)
Acronym: KIDCARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jane C. Burns MD, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 170064
Record Dates: First submitted 2017-01-17; First posted 2017-02-27 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-08

CONDITIONS: Mucocutaneous Lymph Node Syndrome
Keywords: Kawasaki disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Immunoglobulins, Intravenous; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IVIG (Active Comparator): Patient will be randomly assigned to receive a second IVIG infusion: 2 g/kg IV over 8-10 hours single infusion
  Interventions: Drug: IVIG
- Infliximab (Active Comparator): Patient will be randomly assigned to receive Infliximab 10 mg/kg IV over 2 hours
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: IVIG — Subjects randomized to this arm will receive IVIG 2g/kg over 10-12 hours
  Other Names: Intravenous immunoglobulin
  Arms: IVIG
Drug: Infliximab — Subjects randomized to this arm will receive infliximab 10 mg/kg over 2 hours
  Other Names: Remicade
  Arms: Infliximab

SUMMARY:
Kawasaki disease (KD) is a self-limited illness that affects the heart blood vessels (coronary arteries) of infants and children and is now the most common cause of acquired heart disease in children. A mixture of proteins from human blood (Intravenous immunoglobulin, IVIG) is a treatment that reduces the rate of the major complication of the disease: a bulging of the wall of the coronary arteries called an aneurysm. However, 10-20% of children are resistant to this treatment and the fever returns. These children have the highest rates of aneurysm formation and thus should be treated aggressively. Unfortunately, there are no guidelines for the best secondary treatment for these resistant patients because the problem has never been adequately studied. Most physicians choose either a second infusion of IVIG or an engineered antibody called infliximab that inactivates a molecule that promotes inflammation. This trial will randomize (assign by chance like the flip of a coin) IVIG-resistant patients to receive either a second IVIG infusion or infliximab and the response to treatment will be compared to learn which treatment stops the fever the fastest. In addition, parents and caregivers will provide observations about their child's response to the different treatments.

DETAILED DESCRIPTION:
This is a 3-year (2.75-years of enrollment), Phase III, two-arm, randomized, multi-center, superiority treatment study to compare infliximab to a second intravenous immunoglobulin (IVIG) infusion for treatment of persistent or recrudescent fever in children with KD who fail to become afebrile after the first IVIG infusion.

1. Specific aim 1 will test the hypothesis that infliximab will be superior to a second intravenous immunoglobulin (IVIG) infusion for treatment of persistent or recrudescent fever in children with KD who fail to become afebrile after the first IVIG infusion (resistant KD). Cessation of fever (<38°C rectally or orally) within 24h of initiation of study treatment infusion will be the primary outcome measure.
2. Specific aim 2 will test the hypothesis that infliximab treatment will result in more rapid resolution of inflammation compared to second IVIG as measured by the change in white blood cell count (WBC), absolute neutrophil count (ANC), and high-sensitivity C-reactive protein (hsCRP) concentration between baseline and 24 hours and 2 weeks following study treatment.
3. Specific aim 3 will test the hypothesis that infliximab treatment will result in a reduction from baseline in coronary artery Zworst score of ≥ 0.05 standard deviation units as compared to second IVIG at 2 weeks following study treatment measured by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be as follows:

  1. 4 weeks to 17 years of age,
  2. fulfill the American Heart Association case definition for complete or incomplete KD,
  3. have had fever (T ≥38°C) for 3 to 10 days prior to initial IVIG treatment,
  4. have fever (T ≥38°C orally or rectally) between 36 hours and 7 days after end of the first IVIG infusion without other likely cause

Exclusion Criteria:

1. Patient treated with infliximab or steroids for present illness (pts who received oral steroids as outpatients prior to KD diagnosis but who otherwise qualify for the study will not be excluded)
2. Known prior infection with tuberculosis, coccidiomycosis, or histoplasmosis.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane C Burns, MD, Principal Investigator — UCSD
Locations (29):
- United States (29):
  - UAB Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - Memorial Care, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Harbor-UCLA Medical Center, Los Angeles, California
  - UCSF Benioff Children's Hospital-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospital-San Francisco, San Francisco, California
  - Cedar-Sinai Medical Center, West Hollywood, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Health SYstem, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Comer Children's Hospital, Chicago, Illinois
  - Riley Children's Health Indiana University School of Medicine, Indianapolis, Indiana
  - Boston Children's hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Mercy Kansas Ciry, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Maria Fareri Children's Hospital, Valhalla, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of South Dakota Sanford School of Medicine, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Care University of Utah, Salt Lake City, Utah
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burns JC, Roberts SC, Tremoulet AH, He F, Printz BF, Ashouri N, Jain SS, Michalik DE, Sharma K, Truong DT, Wood JB, Kim KK, Jain S; KIDCARE Multicenter Study Group. Infliximab versus second intravenous immunoglobulin for treatment of resistant Kawasaki disease in the USA (KIDCARE): a randomised, multicentre comparative effectiveness trial. Lancet Child Adolesc Health. 2021 Dec;5(12):852-861. doi: 10.1016/S2352-4642(21)00270-4. Epub 2021 Oct 27. PMID 34715057

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVIG | Infliximab
Started | 50 | 55
Participants Who Failed 1st Treatment and Crossed Over to Receive Other Treatment | 22 | 9
Completed | 47 | 51
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Diagnosed with a different disease | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVIG | Infliximab | Total
Number analyzed (Participants) | 49 | 54 | 103
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.1 [1.7 to 5.0] | 3.6 [2.0 to 6.4] | 2.9 [1.7 to 6.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 30 | 29 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 17 | 29
  Not Hispanic or Latino | 36 | 35 | 71
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 6 | 11
  Black or African American | 9 | 10 | 19
  White | 31 | 29 | 60
  Other | 0 | 1 | 1
  Multi-race | 3 | 6 | 9
  Unknown | 1 | 2 | 3
WBC(white blood cells count) [Median (Inter-Quartile Range); unit: cells*10^9/L] | 13.6 [10.7 to 19.2] | 12.8 [8.5 to 16.7] | 13.0 [9.2 to 17.9]
Z-Worst [Median (Inter-Quartile Range); unit: Standard Deviation units] — Z-Worst defined as the greatest internal diameter of the right or left anterior descending coronary artery normalized for body surface area. A Z-score >= 2.5 is considered a aneurysm according to the American Heart Association criteria.
  Standard Deviation units | 1.3 [0.8 to 2.1] | 1.1 [0.7 to 1.7] | 1.3 [0.7 to 1.8]
Illness Day at first IVIG [Median (Inter-Quartile Range); unit: days] — Illness Day at first IVIG treatment for KD, before enrollment into the study
  days | 6.0 [5.0 to 8.0] | 6.0 [5.0 to 7.0] | 6.0 [5.0 to 7.0]
Incomplete KD [Count of Participants; unit: Participants] — Meets 2017 AHA criteria for incomplete KD
  Participants | 15 | 11 | 26
ANC (absolute neutrophil count [Median (Inter-Quartile Range); unit: cells] | 9384.0 [6865.5 to 12752.5] | 8449.0 [5551.5 to 12160.9] | 9062.0 [6062.0 to 12774.0]
zHgb [Median (Inter-Quartile Range); unit: g/dL] — Hemoglobin concentration normalized for age;
  g/dL | -2.3 [-3.5 to -1.4] | -2.3 [-3.0 to -1.3] | -2.3 [-3.1 to -1.3]
PLT (platelet count) [Median (Inter-Quartile Range); unit: cells*10^9/L] | 359.5 [275.8 to 532.8] | 342.0 [241.0 to 398.0] | 349.0 [256.0 to 431.0]
ESR (erythrocyte sedimentation rate), [Median (Inter-Quartile Range); unit: mm/h] | 68.5 [44.8 to 89.3] | 56.5 [41.3 to 86.3] | 63.0 [44.0 to 87.5]
CRP (C-reactive protein) [Median (Inter-Quartile Range); unit: mg/dL] | 9.0 [5.1 to 17.3] | 14.1 [5.9 to 20.1] | 12.0 [5.6 to 20.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cessation of Fever Within 24h of Initiation of Study Treatment With no Fever Recurrence Within Next 7 Days.
Description: A fever will be considered ≥38°C rectally or orally and ≥ 37.5°C axillary. Cessation of fever within 24h of initiation of study treatment with no fever recurrence within next 7 days.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG | Infliximab
Number analyzed (Participants) | 49 | 52
Participants | 25 | 40

2. Secondary Outcome: Change in White Blood Cell Count (WBC) Between Baseline and 24 Hours and 2 Weeks Following Study Treatment.
Description: Change in white blood cell count (WBC), between baseline and 24 hours and 2 weeks following study treatment.
Time Frame: 24h
Measure: Median (Inter-Quartile Range); unit: cells* 10^9/L
Arm/Group | IVIG | Infliximab
Number analyzed (Participants) | 48 | 52
cells* 10^9/L
  Change WBC (Baseline & 24 hr after study treatment completion) | -2.05 [-6.03 to 2.85] | 0.15 [-2.43 to 4.6]
  Change WBC (Baseline & Follow-up Visit ) | -4.9 [-9.7 to 13.4] | -3.5 [-7.7 to 1.25]

3. Secondary Outcome: Change in Zworst Score Between Baseline and 2-week (± 4 Days) Echocardiograms
Description: Zworst score is defined as the largest internal diameter of either the right coronary or left anterior descending arteries normalized for body surface area and expressed as standard deviation units from the mean. A Z-score >= 2.5 is considered a aneurysm according to the American Heart Association criteria.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: Standard Deviation units
Arm/Group | IVIG | Infliximab
Number analyzed (Participants) | 45 | 45
Standard Deviation units | -0.31 [-0.81 to 0.06] | -0.01 [-0.42 to 0.68]

4. Secondary Outcome: Total Number of Fever Days (24 Hour Period With a T≥38.0°C) From Enrollment
Description: Determine the number of days a participant had a fever once the participant has been enrolled into the study.
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | IVIG | Infliximab
Number analyzed (Participants) | 48 | 52
days | 2 [1 to 3.3] | 1 [1 to 2]

5. Secondary Outcome: Duration of Hospitalization
Description: How long a participant was hospitalized for.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | IVIG | Infliximab
Number analyzed (Participants) | 48 | 25
days | 4 [3 to 6] | 2.5 [2 to 4]

6. Secondary Outcome: Number of Participants With IVIG and Infliximab Infusion Reactions and Complications
Description: Determine any complications and/or reactions to each treatment.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | IVIG | Infliximab
Number analyzed (Participants) | 49 | 54
Participants | 1 | 2

7. Secondary Outcome: Change in Absolute Neutrophil Count (ANC) Between Baseline and 24 Hours and 2 Weeks Following Study Treatment.
Description: Change in absolute neutrophil count (ANC) between baseline and 24 hours and 2 weeks following study treatment.
Time Frame: 24h
Measure: Median (Inter-Quartile Range); unit: cells
Arm/Group | IVIG | Infliximab
Number analyzed (Participants) | 48 | 52
cells
  Change ANC (Baseline & 24 hr after study treatment completion | -3398.4 [-7598.45 to 2320.5] | -1742 [-4406.4 to 507.0]
  Change ANC(Baseline & Follow-up visit) | -5853.5 [-10669.6 to -3236.6] | -4661.0 [-8799.3 to -2731]

8. Secondary Outcome: Change in C-reactive Protein (CRP, mg/dL) Concentration Between Baseline and 24 Hours and 2 Weeks Following Study Treatment.
Description: Change in C-reactive protein (CRP, mg/dL) concentration between baseline and 24 hours and 2 weeks following study treatment.
Time Frame: 24h
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | IVIG | Infliximab
Number analyzed (Participants) | 48 | 52
mg/dL
  Change CRP (Baseline & 24 hr after study treatment completion ) | -4.6 [-11.6 to -1.9] | -4.7 [-11.3 to -2.0]
  Change CRP(Baseline & Follow-up visit) | -8.6 [-15.9 to -4.7] | -13.4 [-19.5 to -5.4]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the entirety of the study participation which was 6 weeks from study enrollment.
Arm/Group | IVIG | Infliximab
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/54
Serious Adverse Events (participants affected / at risk) | 27/49 | 10/54
Other Adverse Events (participants affected / at risk) | 6/49 | 14/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IVIG (N=49) | Infliximab (N=54)
Hemolytic Anemia (Blood and lymphatic system disorders) | 10 | 1
Continued Fever after treatment completion and crossover to other study treatment (General disorders) | 22 | 9
Fever following crossover treatment (General disorders) | 3 | 8
Dress Syndrome (Immune system disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IVIG (N=49) | Infliximab (N=54)
GI Symptoms (Gastrointestinal disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Arthritis/pain and swelling in extremities (Musculoskeletal and connective tissue disorders) | 4 | 2
Epistaxis (Blood and lymphatic system disorders) | 3 | 2
Fever after discharge not attributed to KD (General disorders) | 3 | 8
Headache (General disorders) | 2 | 1
URI (Infections and infestations) | 2 | 1
Leukemoid Reaction (Blood and lymphatic system disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Hyperhidrosis (General disorders) | 0 | 1
Pain (IV Site) (Skin and subcutaneous tissue disorders) | 0 | 1
Color Blindness (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03065244/Prot_SAP_000.pdf